CLINICAL TRIAL: NCT04803539
Title: A Prospective, Phase II Trial Using ctDNA to Initiate Post-operation Boost Therapy After Adjuvant Chemotherapy in TNBC (Artemis)
Brief Title: A Prospective, Phase II Trial Using ctDNA to Initiate Post-operation Boost Therapy After Adjuvant Chemotherapy in TNBC
Acronym: Artemis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Liu Qiang, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SunYatsenU2H-LQ4
Record Dates: First submitted 2021-03-16; First posted 2021-03-17 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: stage II-III
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine (Active Comparator): Patients assigned to this group will receive oral capecitabine at a dose of 650 mg/m2 twice a day by mouth for 1 year
  Interventions: Drug: capecitabine
- Capecitabine + Apatinib + Camrelizumab (Experimental): Patients assigned to this group will receive oral capecitabine at a dose of 650 mg/m2 twice a day, Camrelizumab 200mg intravenously, once every two weeks (Q2W), oral apatinib, 250mg, PO, qd for 1 year
  Interventions: Drug: capecitabine + camrelizumab + apatinib

INTERVENTIONS:
Drug: capecitabine — capecitabine is proved to improve 5-year disease-free survival among women with early-stage triple-negative breast cancer who received standard adjuvant treatment(The SYSUCC-001 Randomized Clinical Trial)
  Arms: Capecitabine
Drug: capecitabine + camrelizumab + apatinib — Camrelizumab combined with apatinib is a safe and effective combination proved in patients with advanced TNBC in our early study
  Arms: Capecitabine + Apatinib + Camrelizumab

SUMMARY:
Circulating tumor DNA (ctDNA) has been demonstrated to be an effective prognostic marker in breast cancer. Various studies have shown that early TNBC breast cancer patients with positive ctDNA have high risk of cancer recurrence and worse prognosis. This study aimed to identify TNBC patients with positive ctDNA and initiate boost therapy in these high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years-old at the time of consent to participate this trial
* Stage II - III primary triple negative breast cancer patients(TNBC), TNBC is defined as ER <=1%, PR <=1%；HER2 receptor IHC=1, or IHC=2 and FISH negative.
* positive ctDNA after curative surgery and/or adjuvant chemotherapy
* ECOG 0-2
* If indicated, patient agree to receive adjuvant radiotherapy according to the institutional guidelines
* Patient receives adjuvant chemotherapy according to the NCCN guidelines
* Patient has available tumor tissue from the surgical specimen for next generation sequencing(NCS)
* Patient agrees to give blood samples for ctDNA tests every 3 months in 5 years

Exclusion Criteria:

* Patient has previously received any PD1/PDL1 blockage treatment
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the trial
* Patient with distant metastases of breast cancer beyond regional lymph nodes (stage IV according to AJCC 8th edition)
* Patient participates another interventional clinical trial
* Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 3 years before randomization
* Patient with autoimmune disease preventing the use of camrelizumab
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease Free Survival(IDFS) | 60 months
  Invasive Disease-Free Survival for capecitabine versus capecitabine + apatinib + camrelizumab in ctDNA-positive stage II-III TNBC patients, using STEEP criteria

SECONDARY OUTCOMES:
Distant disease-free survival(DDFS) | 60 months
  Distant Disease-Free Survival for capecitabine versus capecitabine + apatinib + camrelizumab in ctDNA-positive stage II-III TNBC patients, using STEEP criteria
Overall Survival | 60 months
  Overall Survival for capecitabine versus capecitabine + apatinib + camrelizumab in ctDNA-positive stage II-III TNBC patients, using STEEP criteria
Brain metastasis rate | 60 months
  Brain metastasis rate for capecitabine versus capecitabine + apatinib + camrelizumab in ctDNA-positive stage II-III TNBC patients, using STEEP criteria
The rate of adverse effects(AEs) | 60 months
  AEs related to apatinib and/or camrelizumab

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, PhD, Principal Investigator — Sunyat-sen Memorial Hospital
Locations (1):
- Sunyat-sen Memorial Hospital, Guandong, Guangdong, China